CLINICAL TRIAL: NCT07338422
Title: Nonrandomized Controlled Study of HLA-Haploidentical Hematopoietic Stem Cell Transplantation Versus Immunosuppressive Therapy as First-Line Treatment for Severe Aplastic Anemia
Brief Title: HID-HSCT Versus IST as First-line Treatment for SAA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025089
Record Dates: First submitted 2025-09-25; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Aplastic Anaemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HID-HSCT (Experimental)
  Interventions: Procedure: tranplantation
- IST (Other)
  Interventions: Procedure: IST (ATG + CsA+TPORA)

INTERVENTIONS:
Procedure: IST (ATG + CsA+TPORA) — The selection of treatment regimens for subjects is based on clinical decision-making in real-world practice, comprehensively considering factors including patient age, donor matching status, comorbidities, and treatment preferences, with non-randomized group allocation.
  Patients in the immunosuppressive therapy group receive a regimen comprising anti-thymocyte globulin (ATG) + cyclosporine A (CSA) + thrombopoietin receptor agonist (TPO-RA).
  Arms: IST
Procedure: tranplantation — The selection of treatment regimens for subjects is based on clinical decision-making in real-world practice, comprehensively considering factors including patient age, donor matching status, comorbidities, and treatment preferences, with non-randomized group allocation.
  Patients in the transplantation group undergo haploidentical hematopoietic stem cell transplantation (haplo-HSCT).
  Arms: HID-HSCT

SUMMARY:
This study aims to compare the efficacy and safety of HLA-haploidentical hematopoietic stem cell transplantation (HLA-haplo HSCT) versus optimal immunosuppressive therapy (IST) as first-line treatments for severe aplastic anemia (SAA) through a real-world cohort design. The selection of treatment regimens for subjects is based on clinical decision-making in real-world practice, comprehensively considering factors including patient age, donor matching status, comorbidities, and treatment preferences, with non-randomized group allocation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Confirmed diagnosis of severe aplastic anemia, including very severe aplastic anemia, severe aplastic anemia, and hepatitis-associated severe aplastic anemia.

  (2) Age 14-70 years. (3) No HLA-matched related donor available. (4) HIV negative, HBV negative, HCV negative. (5) No absolute contraindications to transplantation or immunosuppressive therapy.

  (6) Signed informed consent form must be obtained before study procedures begin; for subjects aged 18 years or older, informed consent shall be signed by the patient themselves or direct family members. Considering the patient's medical condition, if the patient's own signature is medically inadvisable, the informed consent shall be signed by a legal guardian or the patient's direct family member.

Exclusion Criteria:

1. Inherited bone marrow failure syndromes (IBMFS), including Fanconi anemia, dyskeratosis congenita, Shwachman-Diamond syndrome (SDS), etc.;
2. Clonal cytogenetic abnormalities or bone marrow examination suggesting pre-MDS or MDS;
3. Known severe allergy to ATG;
4. Previous allogeneic or autologous hematopoietic stem cell transplantation;
5. Previous solid organ transplantation;
6. Uncontrolled infection at enrollment, or requiring mechanical ventilation or hemodynamic instability;
7. Active HIV replication at enrollment, detectable HCV antibody positivity and HCV-RNA positivity within 90 days prior to enrollment, or HBsAg positivity; known seropositivity for HIV or active hepatitis C virus;
8. History of malignant tumors (except resected basal cell carcinoma or treated cervical carcinoma in situ);
9. Psychiatric disorders or other conditions that prevent compliance with study treatment and monitoring requirements;
10. Inability or unwillingness to sign the consent form;
11. Other special circumstances deemed ineligible by the investigator.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2030-09-14 (Estimated); Study Completion 2030-09-14 (Estimated)

PRIMARY OUTCOMES:
Failure Free Survival, FFS | 2 year
  survival with complete response whereas death, graft failure and relapse are considered treatment failures

SECONDARY OUTCOMES:
Overall Survival, OS | 2 year
Treatment Related Mortality, TRM | 2 year
  Transplantation-related mortality (TRM) was defined as death without graft failure
hematology remission | 2 year
  hematology recovery, including WBC, Hb and PLT
Infection incidence | 2 year
GVHD incidence | 2 year
QoL evaluation | 2 year
  life quality assessment

IPD SHARING:
Plan to Share IPD: No